CLINICAL TRIAL: NCT04710329
Title: High-Dose Vitamin C Treatment in Critically Ill COVID-19 Patients, A Retrospective Cohort Study
Brief Title: High-Dose Vitamin C Treatment in Critically Ill COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, nurcan coskun, specialist medical doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: CVIT-3334
Record Dates: First submitted 2021-01-13; First posted 2021-01-14 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Respiratory Distress Syndrome, Adult; Covid19
Keywords: coronavirus disease 2019; Ascorbic Acid; intensive care
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19 | interventions — Ascorbic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- C Vit: The patients who were admitted to the intensive care unit and received a high dose intravenous vitamin C protocol constituted the treatment group
  Interventions: Drug: Ascorbic acid
- non-C Vit: The patients who were admitted to the intensive care unit but did not receive the vitamin C protocol constituted the control group
  Interventions: Drug: Ascorbic acid

INTERVENTIONS:
Drug: Ascorbic acid — The daily administration of 6 grams of vitamin C intravenously in 4 equal doses every 6 hours occurred and the treatment lasted 96 hours. Vials containing 1.5 gr vitamin C were placed in 100 cc 5% dextrose and infused intravenously in 30-60 minutes. Prepared serum bottles and sets are wrapped with aluminum foil in order to protect them from sunlight.

SUMMARY:
Acute respiratory failure due to COVİD-19 pneumonia has poor prognosis and high mortality . Both the lack of an effective antiviral treatment and the low level evidence of the recommendations presented in the guidelines on other treatment methods have highlighted supportive treatments. Studies suggest that high-dose vitamin C treatment reduces mortality in patients with sepsis and ARDS, and may also be beneficial in COVİD-19 disease. In the study; the investigator aimed to determine the effect of Vitamin C on short-term mortality and length of intensive care stay in COVID-19 patients.

DETAILED DESCRIPTION:
SARS-CoV-2 causes tissue damage in the endothelium and epithelium, increased vascular permeability and increased plasma levels of IL-6, IL-2, IL-7, IL-10 causing interstitial fibrosis in the lung is considered. Considering these factors in pathogenesis, a picture with high mortality from acute respiratory failure to severe ARDS emerges in critically ill COVID-19 patients. However, despite numerous studies, an effective antiviral treatment has not yet been found in COVID-19 disease. The low level of evidence for the recommendations presented in the guidelines on both treatment and mechanical ventilation has brought supportive treatments to the agenda. Recently, many articles have been published on the potential effects of anti-inflammatory and antioxidant treatments such as high-dose vitamin C, vitamin D, zinc and ozone therapy. In particular, high-dose intravenous vitamin C treatment is inexpensive, easily accessible, and it reduces mortality in patients with sepsis and ARDS in studies, suggesting that it may be beneficial in COVID-19 disease. this is a retrospective cohort study. The main goal of the study; to compare patients who did not receive high-dose vitamin C treatment in the first period of the epidemic and those who received treatment in the next period. the investigator aimed to determine the effect of Vitamin C on short-term mortality and length of stay in intensive care in critically ill COVID-19 patients. All patients' data on age, gender, body mass index, comorbidities (diabetes mellitus, hypertension, coronary artery disease, chronic obstructive pulmonary disease, other), PaO2 / FiO2 ratios, SOFA scores, ferritin, C-Reactive Protein, procalcitonin, lactate, neutrophil and lymphocyte values will be collected by scanning the hospital information system.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with diagnosis of COVID-19, diagnosis confirmed by PCR test
* pneumonia due to COVID-19 was diagnosed with clinical and radiological findings
* Patients who developed acute respiratory failure (PaO2 / FiO2 300 despite the use of 6 l / min reservoir mask) caused by COVID-19 pneumonia
* Older than 18 year

Exclusion Criteria:

* Renal failure
* Hepatic failure
* End-stage malignity
* Primary lung disease (lung cancer, cardio-pulmonary edema)
* Patients who treated with tocilizumab
* Presence of diabetic ketoacidosis, use of insulin infusion, or frequent need for point-of-care glucose monitoring (>6 times/24 hour period) as determined by treating physician
* Active kidney stone
* patients with hospitalization in ICU less than 96 hours

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who admitted to the intensive care unit with the diagnosis of acute respiratory failure due to COVID-19 pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
short term mortality | days 1-28
  Incidence of mortality at 28 days by all causes
Length of Intensive Care Unit Stay | up to 28 days
  Length of Intensive Care Unit Stay

SECONDARY OUTCOMES:
vasopressor requirement | 1-28 days
  all types of vasopressor requirement in intensive care stay
invasive mechanical ventilation requirement | 1-28 days
  invasive mechanical ventilation requirement
PaO2/FiO2 ratio | 1-4 day
  Change in PaO2/FiO2 ratio from admission to 4th day
C-reactive protein | 1-4 days
  Change in C-reactive protein from admission to 4th day
procalcitonin | 1-4 days
  Change in procalcitonin from admission to 4th day
Lymphocyte count | 1-4 days
  Change in Lymphocyte count from admission to 4th day
ferritin | 1-4 days
  Change in ferritin from admission to 4th day
SOFA | 1-4 days
  Change in Sequential Organ Failure Assessment score from admission to 4th day.

CONTACTS AND LOCATIONS:
Overall Officials: Surhan Çınar, Study Chair — Sisli etflal resource and training hospital
Locations (1):
- Sisli etfal training and resource hospital, Şişli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fowler AA 3rd, Truwit JD, Hite RD, Morris PE, DeWilde C, Priday A, Fisher B, Thacker LR 2nd, Natarajan R, Brophy DF, Sculthorpe R, Nanchal R, Syed A, Sturgill J, Martin GS, Sevransky J, Kashiouris M, Hamman S, Egan KF, Hastings A, Spencer W, Tench S, Mehkri O, Bindas J, Duggal A, Graf J, Zellner S, Yanny L, McPolin C, Hollrith T, Kramer D, Ojielo C, Damm T, Cassity E, Wieliczko A, Halquist M. Effect of Vitamin C Infusion on Organ Failure and Biomarkers of Inflammation and Vascular Injury in Patients With Sepsis and Severe Acute Respiratory Failure: The CITRIS-ALI Randomized Clinical Trial. JAMA. 2019 Oct 1;322(13):1261-1270. doi: 10.1001/jama.2019.11825. PMID 31573637
- [Background] Fowler AA 3rd, Fisher BJ, Kashiouris MG. Vitamin C for Sepsis and Acute Respiratory Failure-Reply. JAMA. 2020 Feb 25;323(8):792-793. doi: 10.1001/jama.2019.21987. No abstract available. PMID 32096845
- [Background] Kim WY, Jo EJ, Eom JS, Mok J, Kim MH, Kim KU, Park HK, Lee MK, Lee K. Combined vitamin C, hydrocortisone, and thiamine therapy for patients with severe pneumonia who were admitted to the intensive care unit: Propensity score-based analysis of a before-after cohort study. J Crit Care. 2018 Oct;47:211-218. doi: 10.1016/j.jcrc.2018.07.004. Epub 2018 Jul 5. PMID 30029205
- [Background] Moskowitz A, Huang DT, Hou PC, Gong J, Doshi PB, Grossestreuer AV, Andersen LW, Ngo L, Sherwin RL, Berg KM, Chase M, Cocchi MN, McCannon JB, Hershey M, Hilewitz A, Korotun M, Becker LB, Otero RM, Uduman J, Sen A, Donnino MW; ACTS Clinical Trial Investigators. Effect of Ascorbic Acid, Corticosteroids, and Thiamine on Organ Injury in Septic Shock: The ACTS Randomized Clinical Trial. JAMA. 2020 Aug 18;324(7):642-650. doi: 10.1001/jama.2020.11946. PMID 32809003